CLINICAL TRIAL: NCT05975385
Title: Acupuncture For Prevention Of Postoperative Nausea And Vomiting In Patients Undergoing Laparoscopic Cholecystectomy - A Randomized Controlled Trial
Brief Title: Acupuncture for Prevention of Postoperative Nausea and Vomiting After Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Jaime Ortiz, Professor of Anesthesiology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-53767
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Cholecystitis, Acute; Cholelithiasis; Nausea, Postoperative; Vomiting, Postoperative; Pain, Postoperative
MeSH Terms: conditions — Cholecystitis, Acute; Cholelithiasis; Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. Group 1 - Acupuncture Group 2 - No acupuncture
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient will be under general anesthesia when treatment provided. They will not know whether or not they received acupuncture treatment. Postoperative assessors will not know which group the patient is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Acupuncture (Experimental): Group Acupuncture: Points PC 6 bilaterally, LI 4 bilaterally, and Yin Tang will be needled using Seirin L Type 0.25 X 40 mm needles. MH 6 is located 2 cun (a traditional Chinese unit of length) above the wrist crease in between the tendons of palmaris longus and flexor carpi radialis. LI 4 is in the middle of first and second metacarpal bones. Yin Tang is located between the eyebrows. All needles will be removed once skin closure begins, and before emergence and extubation.
  Interventions: Device: Acupuncture
- Control (No Intervention): No acupuncture treatment provided

INTERVENTIONS:
Device: Acupuncture — Acupuncture at points points PC 6 bilaterally, LI 4 bilaterally, and Yin Tang
  Arms: Acupuncture

SUMMARY:
The purpose is to find out if intraoperative acupuncture performed by needling PC 6 and LI4 point bilaterally, and Yin Tang point will help reduce the incidence postoperative nausea and vomiting in patients undergoing laparoscopic cholecystectomy when added to a prophylactic regimen consisting of ondansetron and dexamethasone. The hypothesis is that the addition of this acupuncture treatment to ondansetron and dexamethasone given for prophylaxis will help reduce the incidence of postoperative nausea and vomiting in patients undergoing laparoscopic cholecystectomy when compared to patients receiving ondansetron and dexamethasone without acupuncture.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ages 18-64
2. American Society of Anesthesiology Physical Status I, II or III
3. Patients scheduled to undergo laparoscopic cholecystectomy at Harris Health System Ben Taub Hospital

Exclusion Criteria:

1. Scheduled open cholecystectomy - excluded due to increased levels of pain in open procedures
2. Renal dysfunction (Serum Cr > 1.2) - excluded due to potential altered metabolism of anesthetic and perioperative medications
3. Allergy to any of the standard anesthetic agents
4. Patient inability to properly communicate with investigators (language barrier, dementia, delirium, psychiatric disorder)
5. Patient or surgeon refusal

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting | Postoperative: 0-1 hours, 1-6 hours, 6-12 hours, 12-24 hours
  Incidence of nausea and vomiting after surgery

SECONDARY OUTCOMES:
Postoperative pain | 24 hours
  Pain on scale 1-10 measured on arrival to PACU, discharge from PACU and at 24 hours post surgery
Total opioids used | 24 hours
  Total opioid given, converted to oral morphine equivalents

CONTACTS AND LOCATIONS:
Locations (1):
- Ben Taub Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No